CLINICAL TRIAL: NCT05130216
Title: A Single-arm Pilot Study of Genicular Nerve Radiofrequency Ablation for Chronic Knee Pain After Total Knee Arthroplasty
Brief Title: Genicular Nerve Radiofrequency Ablation for Chronic Knee Pain After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lucas Anderson, Principle Investigator, University of Utah
Other Study IDs: 144989
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Total Knee Arthroplasty
Keywords: Genicular Nerve Radiofrequency Ablation; Total Knee Arthroplasty; Chronic Knee Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total Knee Arthroplasty: Patients who have undergone total knee arthroplasty post one-year.
  Interventions: Other: Genicular Nerve Radiofrequency Ablation

INTERVENTIONS:
Other: Genicular Nerve Radiofrequency Ablation — Radiofrequency Ablation (RFA)

SUMMARY:
Determine if genicular nerve radiofrequency ablation (RFA) is a clinically effective intervention for patients with chronic knee pain post-total knee arthroplasty (TKA) as defined by pain.

DETAILED DESCRIPTION:
More than 600,000 total knee arthroplasty (TKA) surgeries are performed each year in the United States, and approximately 20% of patients will experience some element of chronic knee pain or dissatisfaction related to pain following this procedure. The options for management are limited, and physicians often resort to chronic opioid management. This creates a less than ideal situation for our elderly population who are more sensitive to the deleterious effects of opioids and who would greatly benefit from pain-free, independent mobility. The investigators propose a single-arm pilot study looking at performing fluoroscopically guided genicular nerve radiofrequency ablation (RFA) for patients with chronic (>6 months) knee pain following a TKA.

A new paradigm for treating post-TKA pain may be the use of RFA of the articular sensory nerve supply of the knee capsule, to desensitize the knee by blocking sensory afferents of the anterior capsule and thereby decreasing pain. While this modality has demonstrated efficacy for chronic knee pain due to osteoarthritis (OA) in the native knee, only one underpowered study has investigated this technique in chronic pain post-TKA. Further, this study targeted only three genicular nerves, while newer cadaveric studies have suggested multiple additional sensory nerves which if ablated may result in increased pain relief. A placebo-controlled explanatory trial of genicular nerve RFA for chronic pain post-TKA of appropriate size and statistical methodology has not been conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 90 years
* At least one year post TKA
* Have no indications for revision TKA
* ≥4/10 knee pain for >6 months following TKA
* ≥80% relief with diagnostic genicular nerve blocks
* Willingness to undergo fluoroscopy-guided genicular nerve RFA treatment.

Exclusion Criteria:

* Conditions that preclude RFA (e.g. pregnancy, pacemaker/ICD, severe cardiac/pulmonary compromise; acute illness/infection; coagulopathy or bleeding disorder; allergic reactions/contraindications to a local anesthetic.
* Inability to write, speak or read in English
* Patient refusal
* Significant psychiatric comorbidity

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have high pain following total knee replacement identified in clinic.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Numeric ranking scale (NRS) pain | Prior to nerve radiofrequency ablation (RFA)
  NRS pain score (0 no pain - 10 severe pain)
Numeric ranking scale (NRS) pain | 1-month post-genicular nerve RFA
  NRS pain score (0 no pain - 10 severe pain)
Numeric ranking scale (NRS) pain | 3-months post-genicular nerve RFA
  NRS pain score (0 no pain - 10 severe pain)
Numeric ranking scale (NRS) pain | 6-months post-genicular nerve RFA
  NRS pain score (0 no pain - 10 severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Anderson, MD, Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No